CLINICAL TRIAL: NCT01696565
Title: PG2 Phase I/II Clinical Study Intravenously Administered in Patients With Advanced Malignancy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PH-CP002-2
Record Dates: First submitted 2011-03-28; First posted 2012-10-01 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Neoplasm Metastasis; Neoplasm Recurrence
Keywords: myelosuppression; chemotherapy; Astragalus membranaceus; hematopoietic response
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 125 mg/day Treatment Arm (Experimental): 125 mg/day PG2 treatment continuously for 7 days
  Interventions: Drug: PG2
- 250 mg/day Treatment Arm (Experimental): 250 mg/day PG2 treatment continuously for 7 days
  Interventions: Drug: PG2
- 500 mg/day Treatment Arm (Experimental): 500 mg/day PG2 treatment continuously for 7 days
  Interventions: Drug: PG2

INTERVENTIONS:
Drug: PG2 — Injectable

SUMMARY:
The objectives of this Phase I/II study are:

1. To find out the maximum tolerated dose (MTD) of PG2 in patients with advanced malignancy receiving chemotherapy and to define a "Study Dose" for Phase II.
2. To evaluate the hematopoietic and immunological responses after administering of PG2. Primarily to study the biological response of PG2, defined as WBC count in this study, and secondarily to study the immunological factors, IL-2, IL-6, TGF-beta, and G-CSF.

DETAILED DESCRIPTION:
This study is the first step for PG2 clinical development in Taiwan in order to further establish its safety and efficacy profile and to build the basis for larger trials.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have malignancy with metastatic or recurrent diseases.
* Patient must have a minimum of thirteen days period elapsed from any previous chemotherapy or radiotherapy and all treatment-related toxicities subsided.
* Patient must have at least 2 courses of chemotherapy treatment left, and a minimum of 13 days between the administration of the last dose of the chemotherapy with PG2 and the start of the next course of chemotherapy.
* Performance status is 0-2 by ECOG scale.
* Patient's compliance and geographic proximity that allow adequate follow up.
* Adequate bone marrow function before the chemotherapy
* Adequate liver and renal function before the chemotherapy
* Written informed consent from patients
* Woman with childbearing potential should use contraception method through the whole PG2 treatment course.
* After the previous course of chemotherapy, the nadir of WBC dropped between 1000 to 3000/ mm3 (for phase II only).

Exclusion Criteria:

* PG2 skin test is positive.
* Active infection
* Breast feeding
* Prior radiotherapy more than 30% of the bone marrow involved.
* Pregnant woman
* Bone marrow transplantation or brain disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2001-12 (Actual); Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Phase I: To find the maximum tolerated dose (MTD) or the highest tolerated dose (HTD) as the study dose of PG2; Phase II: To use the study dose and assess the WBC level of PG2 | within 14 days of each chemotherapy cycle
  For phase I study, the primary endpoint is to determine a safe dosage of PG2 by the dose escalation design.
  For phase II study, the primary endpoint is to compare the WBC level between PG2 plus chemotherapy and chemotherapy alone.

SECONDARY OUTCOMES:
Phase II: To use the study dose to assess the hematopoietic and immunological cytokine levels | within 14 days of each chemotherapy cycle
  For phase II study, the secondary endpoint is to compare the levels of IL-2, IL-6, TGF-beta and G-CSF between PG2 plus chemotherapy and chemotherapy alone.

CONTACTS AND LOCATIONS:
Overall Officials: Woei-Yao Kao, Chief, Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan